CLINICAL TRIAL: NCT04918381
Title: A Multicenter, Prospective, Treat and Resect Feasibility Study of the CellFX System for the Treatment of Low-Risk Basal Cell Carcinoma (BCC) Lesions
Brief Title: CellFX Treat & Resect Low-Risk BCC Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulse Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-TR-014
Record Dates: First submitted 2021-05-30; First posted 2021-06-08 (Actual); Results first posted 2022-12-14 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: BCC - Basal Cell Carcinoma; BCC; Excision Margin
Keywords: CellFX; Nano-Pulse Stimulation; NPS; Clearance
MeSH Terms: conditions — Carcinoma, Basal Cell; Margins of Excision

STUDY DESIGN:
Intervention Model Description: CellFX System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CellFX Procedure (Experimental): Treatment of the BCC with CellFX System
  Interventions: Device: CellFX System

INTERVENTIONS:
Device: CellFX System — Nano-Pulse Stimulation (NPS)

SUMMARY:
This prospective, multicenter, study is designed to evaluate the safety and effectiveness of the CellFX System in adults subjects with low-risk basal cell carcinoma (superficial and nodular) for complete histological clearance of the target lesion followed by surgical tumor excision 60 days post-treatment.

DETAILED DESCRIPTION:
The study will enroll healthy adult subjects with confirmed low-risk (superficial and nodular) BCC lesion(s) by biopsy, excluding BCCs located on the face, neck, scalp, axilla, hands, feet, and genitals not exceeding 1.5 cm. Macrophotography of all study BCCs will be captured and clinically assessed by the site investigator for characterization of healing and scar appearance prior to and post-surgical excision. All subjects will be followed at 3, 7, 14, 30 and 60-days post-CellFX procedure and at 14, 30 and 60-days post-excision. Adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 22 and no older than 85 years of age.
* Subject has 1-2 primary, non-recurrent, superficial, or nodular visible basal cell carcinoma lesion up to 1.5 cm in size with well-defined borders that has been verified by biopsy.
* Lesion(s) is appropriate for full linear excision with 5 mm margins.
* Subject is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Subject gives voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subject is willing to have BCC lesion(s) treated in a single treatment session and must comply with all study procedures including follow-up visits.
* Subject consents to have photographs taken of the BCC lesion(s).
* Subject agrees to refrain from using all other lesion removal products or treatments (topical medication including over-the-counter medications or treatments from PI or another physician) during the study period.
* Subject agrees to refrain from prolonged sun exposure of the treatment area during the study period.

Exclusion Criteria:

* Subject has an implantable electronic medical device (i.e., pacemaker, implantable cardioverter defibrillator).
* Subject has an active infection or history of infection in designated test area within four weeks prior to treatment.
* Subject is not willing or able to sign the Informed Consent.
* Subject is known to be immune compromised/has a history of immunosuppression (e.g., organ transplant, long-term use of psoralen) or genetic disease (e.g., nevoid basal cell carcinoma syndrome [Gorlin syndrome], xeroderma pigmentosum).
* The basal cell carcinoma lesion intended for treatment with the CellFX System is on the face, neck, scalp, axilla, hands, feet, or genitals.
* The basal cell carcinoma intended for treatment with the CellFX System is a high-risk BCC subtype including perineurial, infiltrative, sclerosing, morpheaform, desmoplastic, micronodular, basosquamous or exhibiting aggressive growth patterns.
* Subject is known to be a keloid producer.
* Subject has allergies to Lidocaine or Lidocaine-like products.
* Subject has a history of radiation to the area intended for treatment.
* Subject has current or prior metastatic BCC.
* Subject is currently being treated or has been previously treated with Sonidegib or Vismodegib.
* Subject has recurrent BCC lesions.
* Subject has a systemic infection.
* Subject has a history of epilepsy.
* Subject has a history of cardiac arrhythmia, myocardial infarction or structural heart disease.
* Subject is employed by the sponsor, clinic site, or entity associated with the conduct of the study.
* Subject has any condition or situation which, in the Investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study.
* Subject has a history of use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study, with the exception of participation in a COVID vaccination related clinical trial.

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Nuccitelli, PhD, Study Chair — Pulse Biosciences, Inc.
Locations (5):
- United States (5):
  - Surgical Dermatology Group, Vestavia Hills, Alabama
  - Moy-Fincher-Chipps Dermatology, Beverly Hills, California
  - Palm Harbor Dermatology, Clearwater, Florida
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Clinical Research Center of the Carolinas, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: BCC Lesions
Period: Overall Study
Arm/Group | CellFX Procedure
Started | 30; 37 BCC Lesions
Completed | 30; 37 BCC Lesions
Not Completed | 0; 0 BCC Lesions

BASELINE CHARACTERISTICS:
Population: The total number of enrolled subjects in this study was 30 participants with 37 lesions.
Arm/Group | CellFX Procedure
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Histological presence of superficial or nodular BCC [Number; unit: lesions] | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With BCC Histological Clearance
Description: The primary effectiveness endpoint is the total number of lesions with complete histological clearance of the BCC lesion during histological review of microscopic analysis using H & E slides. Counts and proportions will be assessed.
Time Frame: 60-days post-CellFX procedure
Measure: Count of Units; unit: BCC Lesions
Units Other Than Participants: BCC Lesions
Arm/Group | CellFX Procedure
Number analyzed (Participants) | 30
Number analyzed (BCC Lesions) | 37
BCC Lesions | 34

2. Primary Outcome: Number of Participants With Treatment Related Serious Adverse Events
Description: No serious adverse events related to CellFX Treatment or Procedure
Time Frame: 60-days post-CellFX procedure
Measure: Count of Participants; unit: Participants
Arm/Group | CellFX Procedure
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events were collected during the course of study at Visit days at 0 days, 3 days, 7 days, 14 days, 30 days, and 60 days after CellFX Treatment and at 14 days, 30 days, and 60 days post-surgical excision (total time period of 120 days).
Arm/Group | CellFX Procedure
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CellFX Procedure (N=30)
Folliculitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04918381/Prot_SAP_000.pdf